CLINICAL TRIAL: NCT06586814
Title: A Randomized Study of Suture Versus Staples for Wound Closure in Orthopaedic Trauma Surgery
Brief Title: Suture Versus Staples for Wound Closure in Orthopaedic Trauma Surgery
Acronym: SvS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Joshua Gary, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-24-00012
Record Dates: First submitted 2024-07-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lower Extremity Fracture
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture (Other): Wound Closure
  Interventions: Other: Suture
- Staple (Other): Wound Closure
  Interventions: Other: Staple

INTERVENTIONS:
Other: Suture — Wound Closure
  Arms: Suture
Other: Staple — Wound Closure
  Arms: Staple

SUMMARY:
This pilot study is designed to assess the feasibility of comparing skin closure methods - sutures versus staples - and subsequent rates of surgical site infection following open reduction and internal fixation surgery for orthopaedic trauma injuries. The primary objectives are to determine if enrollment, randomization, and compliance are feasible and to refine data collection methods. Patients =18 years of age with closed fractures of the tibial plateau, tibial pilon, patella, and distal femur presenting within 3 weeks of injury undergoing definitive treatment of their fracture will be approached for participation. If enrolled, they will be randomized to having their surgical wound closed with either nylon sutures or metallic staples. Patient follow up will be standard of care besides answering PROMIS surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients 18-80 years old
* Tibial Pilon, Tibial Plateau Fractures, Patella Fractures, and Distal Femur Fractures
* Incisions must be able to be approximated with subdermal sutures intraoperatively
* English and Spanish speaking patients only

Exclusion Criteria:

* Open fractures
* Incarcerated patients
* Pregnant patients
* Patients who do not speak English or Spanish
* History of infection at surgical incision site at the time of definitive fixation
* Pre-existing skin condition associated with risk of infection (psoriasis, eczema)
* Unable to obtain consent from patient prior to surgery or from legally authorized representative (LAR) prior to skin closure if the patient is unable to consent dur to their medical condition.
* The absence of a subcutaneous closure during the index procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participant enrollment | 12 Months
  - Hitting target enrollment in 12 months, enrolling 50% of eligible patients
Feasibility of randomization to each of the treatments | 6 Months
  - Rate of consent
Assess Protocol Compliance | 6 Months
  * Percentage of survey completion
  * Percentage of follow-up
  * Percentage of completed planned outcomes measures

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No